CLINICAL TRIAL: NCT00145561
Title: The Pharmacokinetics of SAquinavir (Invirase New Tablet Formulation) 1,000mg + Ritonavir (Norvir) 100mg q12h in HIV-infected Pregnant Women (SARA)
Brief Title: The Pharmacokinetic Study of Saquinavir New Tablet Formulation in HIV-infected Pregnant Women.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: D.M. Burger PharmD PhD, hospital pharmacist, Radboud University Nijmegen Medical Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 04.02; MV19059
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2008-10

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Saquinavir and Ritonavir

SUMMARY:
Pharmacokinetic study of Saquinavir and Ritonavir in HIV-infected pregnant women

DETAILED DESCRIPTION:
It is generally accepted that HIV-infected pregnant women should receive treatment to prevent the transmission of HIV from mother-to-child.The (relative) contra-indications for the NNRTIs during pregnancy make a PI based regimen the most rational choice. Based on several experiences and investigations it is expected that saquinavir will play a role as a component of tripe drug regimens for HIV-infected pregnant women. Since the bid dose regimen of 1,000mg saquinavir and 100mg ritonavir is approved by the regulatory authorities and with the availability of a new 500mg tablet formulation of saquinavir,there is a need for a well-designed pharmacokinetic trial using the new 500mg saquinavir tablet formulation in the above mentioned dose.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected woman
* 18 - 40 years of age
* able and willing to sign Informed Consent
* pregnant for a maximum of 31 weeks

Exclusion Criteria:

* history of sensitivity/idiosyncrasy to the drug
* relevant history of interference with drug metabolism
* inability to understand trial procedures
* abnormal specific serum levels
* use of specific concomitant medications
* active hepatobiliary or hepatic disease
* previous failure of saquinavir/ritonavir regimen

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics at week 20 and 33 of gestation and 6 weeks post partum

SECONDARY OUTCOMES:
antiviral activity
safety

CONTACTS AND LOCATIONS:
Overall Officials: David M Burger, Dr, Principal Investigator — Radboud University Medical Center
Locations (10):
- Germany (2):
  - University of Bonn, Bonn
  - University of Cologne, Cologne
- Netherlands (4):
  - Rijnstate Hospital, Arnhem
  - University of Leiden, Leiden
  - Radboud University Medical Centre Nijmegen, Nijmegen
  - Erasmus Medical Centre, Rotterdam
- University Hospital ''Germans Trias i Pujol'', Barcelona, Spain
- Clinic Rajdumri Road Pathumwan, Bangkok, Thailand
- United Kingdom (2):
  - Birmingham Heartlands & Sollihull Hospital, Birmingham
  - Chelsea and Westminster Hospital, London

REFERENCES:
- [Result] van der Lugt J, Colbers A, Molto J, Hawkins D, van der Ende M, Vogel M, Wyen C, Schutz M, Koopmans P, Ruxrungtham K, Richter C, Burger D; SARA study team. The pharmacokinetics, safety and efficacy of boosted saquinavir tablets in HIV type-1-infected pregnant women. Antivir Ther. 2009;14(3):443-50. PMID 19474478
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/19474478/